CLINICAL TRIAL: NCT04028908
Title: Remodelling After Trampoline Fracture in Children
Status: Completed | Type: Observational
Sponsor: Peter Klimek (Other)
Collaborators: Medical Research Council Kantonsspital Aarau, Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Peter Klimek, Principal Investigator, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Other Study IDs: 2015-445; ex15Klimek
Record Dates: First submitted 2019-07-10; First posted 2019-07-23 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Trampoline Fracture; Tibial Fracture
Keywords: ventral tilting of the tibial plateau; anterior tilt angle; proximal tibia epiphyseal plate
MeSH Terms: conditions — Tibial Fractures | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: radiographs in two views of the tibia — The anterior tilt angle of the tibia will be measured by two specialized radiologists according to a specific radiological angle measurement tool (PACS Sectra IDS7TM, Linköping, Sweden).

SUMMARY:
The anterior tilting of the proximal tibia epiphyseal plate is a radiological tool for the diagnosis of suspected trampoline fracture. The tibial fracture leads to a ventral tilting of the tibial Plateau. This study is to document the long-term follow-up of the anterior tilt angle and to verify, if there is an uplift of the tibia plateau with correction of the anterior tilt angle to normal values (= remodelling) in order to guarantee optimal treatment of this rare fracture.

ELIGIBILITY:
Inclusion Criteria:

* trampoline fracture of the proximal lower leg

Exclusion Criteria:

* proximal tibial fractures with unclear etiology

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 2-5 years of life with the diagnosis of a trampoline fracture in the radiographs of the tibia in two views at the Kantonsspital Aarau, Universitätsspital Bern, Universitätskinderspital Zürich, UKBB Universitätsspital Basel, Kantonalspital Luzern.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
anterior tilt angle of the tibia | one year after fracture
  radiological measurement of the anterior tilt angle of the tibia (degree)

SECONDARY OUTCOMES:
difference of anterior tilt angle of the fractured tibia compared with the angle of the healthy tibia | one year after fracture
  difference of anterior tilt angle of the fractured tibia compared with the angle of the healthy tibia (degree)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klimek, Dr. med, Principal Investigator — Kantonsspital Aarau
Locations (2):
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - Universitätsspital Bern, Bern